CLINICAL TRIAL: NCT06968143
Title: Evaluating the Impact of Remote Therapeutic Monitoring on Knee Arthroplasty Recovery
Brief Title: Investigating Patient Satisfaction With Smart Knee Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-0508
Record Dates: First submitted 2025-04-30; First posted 2025-05-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Arthroplasty; Knee Replacement; Knee Replacement Arthroplasty; Knee Osteoarthritis
Keywords: Smart Knee Implant; Total Knee Arthroplasty; Remote Therapeutic Monitoring; Persona IQ
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The patients will be receiving, by their choice, either the smart knee implant, or the standard-of-care total knee arthroplasty. The two groups will have the same pre- and post-operative follow-up, except the smart knee implant group will be able to track their progress through a mobile application and see how they compare in their metrics against others of the same age and gender. Patients in both groups will complete the Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) at their pre-operative, 6-week post-operative, 90-day post-operative, and 1-year post-operative appointments, and will also complete satisfaction surveys at their 6-week post-operative, 90-day post-operative, and 1-year post-operative appointments. The investigators will compare KOOS, JR. scores between the two groups and the investigators will also compare satisfaction scores between the smart knee implant and standard-of-care groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Smart Knee Implant (Experimental): This group will receive the smart knee implant during their arthroplasty and will be able to track their progress according to the smart metrics through a mobile application, and will otherwise have the same standard-of-care as the other arm.
  Interventions: Device: Smart Knee Implant
- Standard-of-Care Knee Arthroplasty (No Intervention): This arm includes patients who are receiving the standard-of-care knee arthroplasty and will have standard follow-up with their surgeons.

INTERVENTIONS:
Device: Smart Knee Implant — An important advancement in objective recovery data occurred when the first ever 'smart' knee implant for remote therapeutic monitoring (RTM) after total knee arthroplasty (TKA) was released in 2021. The implant includes both a prosthesis for TKA and a stem, the latter of which records the following metrics: step count, distance traveled, tibial range-of-motion (ROM), functional ROM, average walking speed, stride length, and cadence. The implant sends the recordings to a mobile platform. Additionally, it collects and analyzes patient across the entire population of users and creates percentiles for each metric based on patient age, gender and time since surgery. These "recovery curves" provide more objective data for practitioners and patients to evaluate recovery progress and make adjustments to their care plans accordingly.
  Other Names: Persona IQ
  Arms: Smart Knee Implant

SUMMARY:
The main goal of this study is to see if there is a connection between the social and economic resources available in a patient's neighborhood (measured by the Area Deprivation Index, ADI) and their recovery after knee replacement surgery, as tracked through remote monitoring. A secondary goal is to find out if patients' self-reported pain and function score are linked to their actual physical improvement after surgery as measured by a remote therapeutic monitoring (RTM) device. Additionally, this study examines whether RTM can reduce the number of postoperative clinic visits within the first 90 days after surgery while maintaining patient satisfaction and patient-reported outcome measures (PROMs).

DETAILED DESCRIPTION:
Predicting and measuring knee function after total knee arthroplasty (TKA) has been a topic of debate in the field of orthopedic surgery for decades. The early recovery period after TKA is a critical time for achieving functional range of motion and mobility. For this reason, patients are traditionally examined at regular intervals during the postoperative period for evaluation. For patients who are not meeting targets during early recovery, interventions such as manipulation under anesthesia (MUA) or modifications to physical therapy protocols can improve outcomes. Remote therapeutic monitoring (RTM) using smart knee implants has been proposed as a means of enhancing postoperative follow-up with increased convenience to patients and without overburdening ambulatory resources. These smart knee implants collect objective recovery data including range-of-motion (ROM), step count, and cadence, and send these metrics to a mobile application so that patients and their practitioners can track their progress outside of the medical space. This study aims to compare post-operative patient-reported outcomes and satisfaction at multiple timepoints between patients with RTM and those with the current standard-of-care.

Insight into patient's functional recovery in their post-operative home environment may help orthopedic surgeons to better understand the impact of the social determinants of health (SDOH) on recovery. One of the methods of quantifying SDOH that has been popular in the healthcare field is the Area Deprivation Index (ADI). ADI was developed by the University of Wisconsin-Madison and uses patient addresses to display percentile-based information about neighborhood resources (including income, education, employment, and housing quality), quantifying healthcare accessibility. Some studies have found that while higher ADI may predict medical complications, non-home discharge, length of stay, and 90-day emergency department visits, there is low to no evidence that the metric is correlated with postoperative readmission rates, reoperation rates, or range of motion (ROM).Therefore, investigation into ADI as a predictor of outcomes following TKA needs to be further studied, particularly in juxtaposition with objective metrics of recovery.

The primary objective of this study is therefore to delineate if there is a correlation between the SDOH resources available to patients based on their home environment as measured by ADI, and remotely monitored functional outcomes after TKA . The secondary objective is to determine if patient-reported pain and function scores as measured by Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) correlate with remotely monitored functional improvement after TKA. The tertiary objective is to determine how patient satisfaction with surgery and postoperative recovery compares between patients with RTM and patients with standard knee replacements.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients undergoing unilateral primary or revision total knee arthroplasty with the smart knee implant or standard-of-care

Exclusion Criteria:

* Patients who receive contralateral knee replacement or contralateral or unilateral hip replacement within 90 days before or after their knee replacement in this study
* Patients with post-operative weight-bearing restrictions or physical deconditioning prohibiting routine physical therapy participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes and Satisfaction | From enrollment to 1 year after arthroplasty
  The patients in both arms will complete surveys on their subjective pain and function as well as their subjective satisfaction with the knee arthroplasty preparation, surgery, and recovery. The investigators will compare these surveys between the experimental group and the standard-of-care group at select time points.

SECONDARY OUTCOMES:
Area Deprivation Index Correlation with Recovery | up to 1 year
  The investigators will be retrospectively collecting patient records that will include patient neighborhood locations to calculate an Area Deprivation Index (ADI) score. These patients will be those who have received the smart knee implant before this study was approved, and the investigators will evaluate the correlation between smart knee implant recovery curve percentiles and the Area Deprivation Index in patients receiving the smart knee implant. A high Area Deprivation Index means being more socioeconomically deprived, and the scale is scored from 0 to 100.
Correlation between Knee Injury and Osteoarthritis Outcome score for Joint Replacement (KOOS, JR.) and smart knee implant recovery curve percentiles | From enrollment to 1 year after arthroplasty
  The investigators will collect the Knee Injury and Osteoarthritis Outcome score for Joint Replacement (KOOS, JR.) and smart knee implant recovery curve percentiles for the patients that receive smart knee implants and will calculate correlation scores between them. The KOOS, JR. is scored from 0 to 100 and a higher score means better knee function.
Complications after Knee Arthroplasty | From enrollment to 1 year after arthroplasty
  The investigators will record the rate of patients requiring assistive walking devices, revision arthroplasty, manipulation under anesthesia, and the rates of periprosthetic joint infection between patients who receive smart knee implants and the standard-of-care joint arthroplasty.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Wallace, MD, Principal Investigator — The University of Chicago Department of Orthopaedic Surgery
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yocum D, Housholder E, Yergler J. Manipulation under Anesthesia Following TKA with Persona IQ: A Case Series. J Orthop Case Rep. 2023 Aug;13(8):127-131. doi: 10.13107/jocr.2023.v13.i08.3844. PMID 37654748
- [Background] Yocum D, Elashoff B, Verta P, Armock G, Yergler J. Patient reported outcomes do not correlate to functional knee recovery and range of motion in total knee arthroplasty. J Orthop. 2023 Jul 27;43:36-40. doi: 10.1016/j.jor.2023.07.009. eCollection 2023 Sep. PMID 37564705
- [Background] Shimizu MR, Buddhiraju A, Lin-Wei Chen T, Huang Z, Chen SF, Xiao P, RezazadehSaatlou M, Kwon YM. Socioeconomic area deprivation index is not associated with postoperative complications following revision total hip and knee joint arthroplasty. J Orthop. 2024 Jul 17;58:135-139. doi: 10.1016/j.jor.2024.07.008. eCollection 2024 Dec. PMID 39100544
- [Background] Calkins FM, Pagani NR, Bragg J, Gauthier Z, Salzler M. Neighborhood socioeconomic disadvantage does not predict need for manipulation under anesthesia or range of motion following total knee arthroplasty. J Orthop. 2024 Jun 15;58:146-149. doi: 10.1016/j.jor.2024.06.013. eCollection 2024 Dec. PMID 39100542
- [Background] Jevnikar BE, Huffman N, Roth A, Klika AK, Deren ME, Zhang C, Piuzzi NS; CCARR Corporate Authorship. Impacts of neighborhood deprivation on septic and aseptic revision total knee arthroplasty outcomes: A comprehensive analysis using the area deprivation index. Knee. 2024 Dec;51:74-83. doi: 10.1016/j.knee.2024.08.006. Epub 2024 Sep 5. PMID 39241673
- [Background] Shimizu MR, Buddhiraju A, Kwon OJ, Kerluku J, Huang Z, Kwon YM. The Utility of Neighborhood Social Vulnerability Indices in Predicting Non-Home Discharge Disposition Following Revision Total Joint Arthroplasty: A Comparison Study. J Arthroplasty. 2025 May;40(5):1148-1153. doi: 10.1016/j.arth.2024.10.118. Epub 2024 Oct 25. PMID 39490785
- [Background] Gordon AM, Ng MK, Elali F, Piuzzi NS, Mont MA. A Nationwide Analysis of the Impact of Socioeconomic Status on Complications and Health Care Utilizations After Total Knee Arthroplasty Using the Area Deprivation Index: Consideration of the Disadvantaged Patient. J Arthroplasty. 2024 Sep;39(9):2166-2172. doi: 10.1016/j.arth.2024.04.028. Epub 2024 Apr 12. PMID 38615971
- [Background] Zimmer Biomet and Canary Medical Announce FDA De Novo Classification Grant and Authorization to Market the World's First and Only Smart Knee Implant n.d. http://investor.zimmerbiomet.com/news-and-events/news/2021/08-30-2021-120155075 (accessed December 12, 2024).
- [Background] Hsu H, Siwiec RM. Knee Arthroplasty(Archived). 2023 Jul 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507914/ PMID 29939691
- [Background] Bourne RB. Measuring tools for functional outcomes in total knee arthroplasty. Clin Orthop Relat Res. 2008 Nov;466(11):2634-8. doi: 10.1007/s11999-008-0468-0. Epub 2008 Sep 9. PMID 18780136
- [Background] Yoshida Y, Zeni J, Snyder-Mackler L. Do patients achieve normal gait patterns 3 years after total knee arthroplasty? J Orthop Sports Phys Ther. 2012 Dec;42(12):1039-49. doi: 10.2519/jospt.2012.3763. Epub 2012 Oct 22. PMID 23090437